CLINICAL TRIAL: NCT03738657
Title: Gustatory Function Following Radiotherapy to the Head and Neck
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR4927
Record Dates: First submitted 2018-08-28; First posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Screening: Olfactory screening
- On Study: Taste testing
  Interventions: Other: Olfactory screening; Other: Quantative Gustatory Testing using Taste Strips

INTERVENTIONS:
Other: Olfactory screening — Therefore prior to gustatory testing, patients will be screened and assessed as having either normal or abnormal olfactory function using the Sniffin' Sticks (Burghart; Wedel, Germany). The test consists of 12 odour pens which represent every-day odours (peppermint, fish, coffee, banana, orange, rose, lemon, pineapple, cinnamon, cloves, leather and liquorice). Patients are presented with an odour and select the perceived smell using a multiple-forced-choice method.
  Groups: On Study
Other: Quantative Gustatory Testing using Taste Strips — Following screening for olfactory function, whole mouth gustatory function will be assessed using validated taste strips (Burghart; Wedel, Germany). Filter paper test strips are impregnated at one end with 2cm2 of either sweet, sour, salty or bitter taste solutions in four concentrations. In a pseudo-randomised sequence, individual strips will be placed on the tongue and patients will be asked to close their mouth in order to assess whole mouth function. Through a forced-choice procedure patients will be asked to identify the taste stimuli. Scores for individual taste qualities will range from 0-4 and an overall taste score will range from 0-16.
  Patients will rinse their mouth with tap water prior the application of each taste strip.
  Groups: On Study

SUMMARY:
The aim of this study is to assess the effect of RT or chemo-RT on chemosensory gustatory function in patients with HNC. By using detailed dosimetric data derived from the RT planning system, we will be able to calculate mean radiation doses to important structures including the anterior and posterior tongue, oral cavity, parotid and submandibular salivary glands, and correlate them with both qualitative and quantitative data for dysgeusia.

DETAILED DESCRIPTION:
This study aims to collect data from patients with HNC undergoing RT or chemo-RT to correlate quantitative chemosensory gustatory function with

* Detailed dosimetric data for critical structures relevant to perception of taste
* Fungiform papillae density (FPD)
* Use of concurrent platinum based therapy
* Patient reported taste loss using The Taste and Smell Survey (TSS) [14]
* Patient reported toxicity and overall QOL using University Washington Quality of Life Revised Version 4 (UW-QOL v4) [15].
* Clinician reported acute and late toxicity using NCI Common Terminology Criteria for Adverse Events Version 4.0 (CTCAE v4) [16] and Scale of Subjective Total Taste Acuity (STTA) [17].
* Weight (as a surrogate of nutritional status).

This study hopes to demonstrate a dose dependent relationship for loss of taste and to develop a dose constraint for preservation of taste. In turn this will serve as a platform for further research to optimise the technical delivery of radiation either in the form of optimised IMRT or through the use of intensity modulated proton therapy (IMPT).

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Undergoing unilateral or bilateral RT or concurrent chemo-RT to the head and neck - region using either a conformal or IMRT planning technique or
* No restrictions on tumour sub-site
* No restriction on tumour histology
* No restrictions on radiotherapy dose and fractionation
* For entry into the cross-sectional cohort; patients 12 months post completion of unilateral or bilateral RT or concurrent chemo-RT to the head and neck region using either a conformal or IMRT planning technique.

Exclusion Criteria:

* Patients with pre-existing olfactory or gustatory disorders either self-reported or through objective taste function testing.
* Patients with radiological or clinical involvement of following nerves

  * facial nerve
  * chorda tympani
  * glossopharyngeal nerve
  * lingual nerve
  * greater petrosal nerve
  * geniculate ganglion
* Patients who have undergone a total or partial glossectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with H&N cancer staged at T1-T4 disease and N0-N3 disease attending RMH who have consented to treatment with curative intent using RT or chemo-RT.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2018-08-29 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
The association between radiotherapy dose and patient-reported dysgeusia at 6 months following RT or chemo-RT for HNC. | At 1 year
  Compare the mean dose delivered to the anterior two thirds of the surface of the tongue for those patients who report clinically significant dysgeusia at 6 months, with those who report clinically insignificant dysgeusia. For the purposes of the primary objective, mean dose (Gy) to the anterior two thirds of the tongue will be used. Patient-reported dysgeusia will be assessed using the Taste and Smell Survey (Q13) and patient results will be dichotomised into clinically significant and clinically insignificant loss of taste.

SECONDARY OUTCOMES:
The association between patient-reported dysgeusia and RT dose to the posterior third of the surface of the tongue, oral cavity, left and right parotid glands, left and right submandibular glands and the use of concomitant chemotherapy. | At 1 year
  patient-reported dysgeusia will be assessed using the Taste and Smell Survey (Q13) and patient results will be dichotomised into clinically significant and clinically insignificant loss of taste as above. dose volume histogram data will generate mean dose to oral cavity structures (including posterior third of tongue, anterior two thirds of the tongue, whole oral cavity, parotid glands, submandibular glands).
The association between RT dose to oral cavity structures and objective dysgeusia | At 1 year
  Through use of using chemosensory testing
The association between either patient-reported dysguesia or objective dysgeusia | At 1 year
  Through using chemosensory testing and the use of concomitant chemotherapy.
The association between patient-reported dysgeusia and percentage change in weight. | At 1 year
  patient-reported dysgeusia will be assessed using the Taste and Smell Survey (Q13) and patient results will be dichotomised into clinically significant and clinically insignificant loss of taste as above.

CONTACTS AND LOCATIONS:
Overall Officials: Chris Prof Nutting, Professor, Principal Investigator — Consultant
Locations (1):
- Head and Neck Unit, Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No